CLINICAL TRIAL: NCT04852744
Title: NEUROIMAGERIE DU TROUBLE DE LA PERSONNALITE BORDERLINE A L'ADOLESCENCE AVEC ET SANS TROUBLE DE STRESS POST-TRAUMATIQUE
Brief Title: NEUROIMAGING OF ADOLESCENT BORDERLINE PERSONALITY DISORDER WITH AND WITHOUT POST-TRAUMATIC STRESS DISORDER
Acronym: BorderStress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: CHU de Rouen - Accueil (Other); Centre Hospitalier Universitaire de Caen (Other); Université de Caen Normandie (Other); Centre Hospitalier du Rouvray (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A00366-51
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Borderline Personality Disorder
Keywords: Adolescence; Hippocampus; Neuropsychology; Borderline personality disorder; Post-traumatic stress disorder
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Borderline girls with PTSD (Other): * female
  * Age between 13 and 17 years inclusive
  * Diagnosis of borderline personality disorder according to the criteria of the Diagnostic and Statistical Manual for mental disorders, fifth edition (DSM-5; American Psychiatric Association, 2013; SIDP-IV)
  * Post-traumatic stress disorder according to DSM-5 criteria (American Psychiatric Association, 2013; K-SADS-PL)
  * Level of general psychopathology compatible with participation in the study (score> 20 on the CGA-S)
  * Oral and written comprehension of the French language
  * Affiliation to the social security scheme
  * Informed consent signed by the legal representatives holding the exercise of parental authority and the adolescent herself
  Interventions: Other: Brain MRI
- Borderline girls without PTSD (Other): * female
  * Age between 13 and 17 years inclusive
  * Diagnosis of borderline personality disorder according to the criteria of the Diagnostic and Statistical Manual for mental disorders, fifth edition (DSM-5; American Psychiatric Association, 2013; SIDP-IV)
  * Level of general psychopathology compatible with participation in the study (score> 20 on the CGA-S)
  * Oral and written comprehension of the French language
  * Affiliation to the social security scheme
  * Informed consent signed by the legal representatives holding the exercise of parental authority and the adolescent herself
  Interventions: Other: Brain MRI
- Healthy controls (Other): * female
  * Age between 13 and 17 years inclusive
  * Absence of mental disorder according to DSM-5 (American Psychiatric Association, 2013 ; K-SADS-PL et SIDP-IV)
  * Oral and written comprehension of the French language
  * Affiliation to the social security scheme
  * Informed consent signed by the legal representatives holding the exercise of parental authority and the adolescent herself
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI — Anatomical MRI The anatomical data will be acquired by means of a 3T Signa Premier General Electric Healthcare MRI, allowing the acquisition of classic anatomical sequences (T1, T2) and a high-resolution hippocampal sequence allowing to accurately apprehend its various sub-fields. (total acquisition time: 10 min).
  The hippocampal volume, the orbital-frontal cortex and the cingulate cortex will be measured by voxel-based morphometry (VBM; Ashburner & Friston, 2000]) using the SPM software (Statistical Parametric Mapping; Friston et al., 2006). The voxel-by-voxel morphometric analysis of T1 MRI images makes it possible to classify and segment the different brain tissues (gray matter versus white matter) and to analyze the focal differences in volume within these tissues between the different groups.
  Other Names: Psychological and behavioural assessment

SUMMARY:
Borderline personality disorder (BPD) is a common mental disorder in adolescents with significant individual and societal repercussions, characterized over the long term by emotional hyperresponsiveness, relational instability, identity disturbances and self-aggressive behavior. The etiology of BPD is multifactorial and involves exposure to traumatic life events, which are present in the majority of cases. This explains the very common co-morbidity between BPD and post-traumatic stress disorder (PTSD), which involves emotionally painful memory relapses of one or more traumatic events, associated with an emotional trauma avoidance syndrome (s). ) and hypervigilance. Brain imaging studies in adolescents with BPD have shown decreases in the volume of gray matter within the frontolimbic network, as well as a decrease in frontolimbic white matter bundles. These brain changes are considered to be biological markers of TPB. However, the exact same brain changes are seen in PTSD. Although it represents more than a third of adolescents hospitalized in psychiatry, neuroscientific studies of BPD in adolescence are still scarce. The expertise we have acquired in U1077 in adolescents with PTSD offers us an exceptional opportunity to characterize in BPD with and without PTSD structural anomalies, including the hippocampus, and functional at rest, never used for hour in the teenager's BPD. Beyond that, carrying out an 18-month follow-up of the patients will allow us to assess the predictive value of these anomalies on the level of general psychopathology in all the patients studied and the intensity of the symptoms of traumatic relapse in the patients with PTSD. This modeling of disorders integrating psychopathological, neuropsychological and neuroanatomical approaches will provide the clinician with new knowledge necessary for therapeutic innovation.

DETAILED DESCRIPTION:
A - RESEARCH OBJECTIVES

1. Primary objective:

   • Compare the hippocampal volume between adolescent girls with BPD with and without PTSD
2. Secondary objectives:

   * 1 - Evaluate the link, transverse and long-term (18 months), between the hippocampal volume and the level of general psychopathology in all the patients studied, and between the hippocampal volume and the intensity of the symptoms of traumatic revival in adolescent girls with PTSD.
   * 2 - Compare the volume of the hippocampal subfields between adolescent girls with BPD with and without PTSD, and assess in patients with PTSD the link, transverse and long-term (18 months), between volumes of the hippocampal sub-fields and intensity symptoms of traumatic revival
   * 3 - Compare the volume and integrity of the white matter bundles of the fronto-limbic network between adolescent girls with BPD with and without PTSD
   * 4 - Compare resting brain activity between adolescent girls with BPD with and without PTSD
   * 5 - Explore the links between changes in the brain and the intensity of the main psychological alterations associated with BPD in adolescence: i) attachment insecurity; ii) emotional dysregulation; iii) attention deficit and dysexecutive syndrome; iv) hypermentalization; and v) autobiographical memory and dissemination of identity.

B - Secondary evaluation criteria:

* 1 - Hippocampal volume (VBM); Global Clinical Assessment Scale score (CGA-S; Endicott et al., 1976); "Réviviscences" score in the French version of the UCLA Post-Traumatic Stress Disorder Reaction Index for Children and Adolescents (UCLA PTSD-RI C / A; Steinberg et al., 2013).
* 2 - Volume of each hippocampal subfield (Ammon's Horn [CA] 1, CA2, CA3, dentate gyrus, subiculum: anatomical MRI; Region Of Interest [ROI] method; Postel et al., 2019); "Intrusion" score of the French version of the UCLA PTSD-RI C / A.
* 3 - Orbitofrontal and cingulate cortex volume (VBM); anisotropy fraction (fractional anisotropy; FA) and average diffusivity (apparent diffusion coefficient; ADC) of fronto-limbic white matter beams (IRM Diffusion Tensor Imaging [DTI]; Le Bihan et al., 2001).
* 4 - Functional connectivity of brain networks in the resting state: default network (default mode network), salience network and central executive network; Viard et al., 2019).
* 5 - Brain modifications (VBM, ROI, AF, ADC, functional connectivity of resting networks) and: i) "Insecure attachment" score to Individual Relationship Model Cards (Ca-MIR; Pierrehumbert et al., 1996); ii) score "Separation-distress" and "Fear" in the French version of the Affective Neuroscience Personality Scale (ANPS; Pahlavan et al., 2008); iii) Continuous Performance Test omission score (CPT; Conners, 2002) and Wisconsin Card Sorting Test perseverance score (WCST; Heaton et al., 1993); iv) "Hypermentalisation" score in the French version of the Movie Assessment of Social Cognition (MASC; Martinez et al., 2017) and of the Reflective Functioning Questionnaire (RFQ; Badoud et al., 2015); and v) measurement of the quality of autobiographical productions (Reese et al., 2011), total score in the French version of the Assessment of Identity Development in Adolescence (AIDA; Goth et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

For the 3 groups:

* female
* Age between 13 and 17 years inclusive
* Oral and written comprehension of the French language
* Affiliation to the social security scheme
* Informed consent signed by the legal representatives holding the exercise of parental authority and the adolescent herself

For patients:

* Diagnosis of borderline personality disorder according to the criteria of the Diagnostic and Statistical Manual for mental disorders, fifth edition (DSM-5; American Psychiatric Association, 2013; SIDP-IV)
* Level of general psychopathology compatible with participation in the study (score> 20 on the CGA-S)

TB + / PTSD + group:

- Post-traumatic stress disorder according to DSM-5 criteria (American Psychiatric Association, 2013; K-SADS-PL)

In the control group :

* Absence of mental disorder according to DSM-5 criteria (American Psychiatric Association, 2013; K-SADS-PL and SIDP-IV)
* Oral and written comprehension of the French language
* Informed consent signed by the legal representative, the holder (s) of the exercise of parental authority and the adolescent herself

Exclusion Criteria:

* - Illiteracy / illiteracy
* Sensory disorder (visual, auditory)
* Severe chronic psychiatric comorbidity: autism spectrum disorder, intellectual disability, schizophrenia spectrum disorder and other psychotic disorders, bipolar disorder
* Severe or current brain pathology (chronic neurological disease, encephalitis, history of severe head trauma), alertness disorder
* History of anoxic coma
* Contraindication to MRI (magnetic foreign body, claustrophobia, contraindication to prolonged lying down)
* Severe physical pathology in progress
* Moving outside the Normandy region planned within 18 months
* The inclusion of the subject in another biomedical research protocol (during the present study)
* Intellectual deficit (IQ <70)
* Pregnant or breastfeeding women

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Hippocampal volume | during the month following inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No